CLINICAL TRIAL: NCT06735768
Title: Double-blind, Randomized, Sham-controlled Study of Closed-loop Repetitive Transcranial Magnet Stimulation (rTMS) for the Short-term Prevention of Migraine
Brief Title: Closed-loop RTMS for Short-term Migraine Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brightmind.AI (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2145/2023
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): This group receives rTMS treatment.
  Interventions: Device: rTMS treatment; Device: Determination of motor hotspot and motor treshold
- Sham group (Sham Comparator): This group receives sham treatment.
  Interventions: Device: Determination of motor hotspot and motor treshold

INTERVENTIONS:
Device: rTMS treatment — Brightmind.AI´s rTMS protocol is applied
  Arms: Active group
Device: Determination of motor hotspot and motor treshold — Determination of motor hotspot and motor treshold

SUMMARY:
Migraine is a prevalent and debilitating primary headache disorder, where patients suffer from disabling symptoms that usually consist of a moderate to severe headache lasting 4 to 72 hours, nausea and/or vomiting, phonophobia and photophobia. Transcranial magnetic stimulation (TMS) is a noninvasive technique that is considered to be safe. Repetitive TMS (rTMS) might be useful for migraine prophylaxis. However, available studies on the use of rTMS for preventive treatment of migraine are limited. Currently, rTMS is not recommended in the recent guidelines for the treatment of migraine published by the German Neurological Society in 2022.

Therefore, the aim of the current study is to provide reliable data on the short-term effect of rTMS for the prevention of migraine. The investigators will follow the Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition, with the exception of study duration, which will be limited to four weeks of baseline, three sessions of rTMS within a 10-day timeframe and 4 weeks of follow-up as our study aims to examine short-term efficacy.

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-65
* Migraine without aura, migraine with aura or chronic migraine according to the diagnostic criteria of the third edition of the International Classification of Headache Disorders (ICHD-3) - Age of onset before 50 years of age
* At least 4 migraine days in each of three subsequent 4- week periods preceding the screening period. (Subsequently, the investigators use month synonymous for 4-week periods)
* At least 4 migraine days during one month of baseline prior to treatment.
* Ability to distinguish migraine headaches from other headache types (e.g., tension-type headaches)
* Willing to adhere to the rTMS regimen and able to monitor MD in Migraine diary
* No changes in medication usage/regime for three months before the start of treatment (incl. use of acute abortion / rescue medication). In case of Erenumab, Fremanezumab, Galcanezumab no changes in usage/regime for six months before the start of treatment. Every medication is reported and documented.
* No changes in medication usage/regime during the entire study period (i.e., keeping acute intervention protocol as previously handled for the past three months; not introducing new approaches in intervention/ prevention during this time period (such as anti-nausea drugs not previously taken)). Every medication is reported & documented.
* Use of a single drug for migraine prophylaxis is permitted as long as the dosage has not been altered within 3 months of starting the study and the dosage must not be altered for the entire duration of the study.
* No other stimulation techniques.
* No change in acupuncture, relaxation training, biofeedback, behavioral therapy or other psychological or psychotherapeutic interventions for three months preceding the study and during the entire study period investigator.
* Ability to read and understand the written information (patient information, migraine diary, CRF and Adverse Events (AE) collecting form)
* Completed baseline headache diary with missing data on not more than 5 of 28 days.

Exclusion criteria:

* More than 26 headache days in any of three subsequent months preceding the screening visit.
* More than 26 headache days during baseline
* Pregnant persons
* Usage of Onabotulinumtoxin A for managing chronic migraines.
* Medication-overuse according to ICHD-3
* Presence of metals or implanted devices that can be in close proximity the of device (i.e., above the neckline) and can be adversely affected by magnetic fields including:

  * Stents
  * Implanted stimulators
  * Implanted vagus nerve or brain implants incl. deep brain stimulators
  * Implanted electrical devices
  * Cochlear implants for hearing
  * Any magnetic implants
  * Bullet fragments
  * Grenade fragments
* Presence of heart pacemakers, defibrillator, intracardiac lines or medication pumps
* Known severe adverse reactions in response to rTMS
* Patients diagnosed with bipolar disorder, substance use disorders or psychosis
* Patients with a known medical history, as well as a family history, of seizures.
* Patients experiencing chronic sleep deprivation
* Patients with structural CNS disorders such as a brain tumor, stroke, or traumatic brain injury.
* Patients with chronic tinnitus in the judgement of the investigator
* Patients with other disorders interfering with the study in the judgement of the investigator.
* Treatment with another investigational drug or other intervention until the end of the study
* Botulinum toxin-based infusions for cosmetic reasons at the forehead within a period of six months prior to study inclusion until the final visit.
* Other clinically relevant pain syndromes
* Depression or anxiety in the judgement of the investigator as assessed by means of BDI-II (score 20 or above) and DASS-21 (score 14 or above).
* Severe health risks in the judgement of the investigator. In particular this includes assessing the risk associated with a history of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Monthly migraine days (MMD) | comparing 4 weeks before with 4 weeks after rTMS
  Mean number of MMD 4 weeks before and 4 weeks after rTMS treatment.

SECONDARY OUTCOMES:
50 percent responder rate | comparing 4 weeks before with 4 weeks after rTMS
  Responder rate as a reduction in MMD by 50 percent or more.
Weekly Migraine days after stimulation. | comparing 4 weeks before with 4 weeks after rTMS
  Mean
Monthly headache days | comparing 4 weeks before with 4 weeks after rTMS
  Mean number of monthly headache days before and after rTMS treatment.
Monthly (4 weeks) days with use of acute medication | comparing 4 weeks before with 4 weeks after rTMS
  Mean number of monthly days with acute medication usage before and after rTMS treatment.
Headache severity | comparing 4 weeks before with 4 weeks after rTMS
  Mean headache severity of migraine headaches before and after rTMS treatment.
Duration of migraine attacks | comparing 4 weeks before with 4 weeks after rTMS
  Mean duration of migraine attacks before and after rTMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wöber, Prof., PhD, Principal Investigator — Medical University Vienna
Locations (1):
- Univ.-Klinik für Neurologie, Medizinische Universität Wien, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No